CLINICAL TRIAL: NCT05083065
Title: Evaluation of Menstrual Irregularities and Abnormal Uterine Bleeding After Covid-19 Vaccine
Acronym: MECOVAC-1
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: MECOVAC-1
Record Dates: First submitted 2021-10-17; First posted 2021-10-19 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: COVID-19; Vaccine; Menstrual Irregularity; Menopausal Bleeding
Keywords: Covid-19 vaccine; Menstrual Irregularity; Menopausal Bleeding
MeSH Terms: conditions — COVID-19; Menstruation Disturbances | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women who underwent Covid-19 vaccination: This group includes women who underwent both the first or complete cycle of Covid-19 vaccination, regardless of the vaccine used.
  Interventions: Biological: Covid-19 vaccine

INTERVENTIONS:
Biological: Covid-19 vaccine — * First dose or complete cycle of Comirnaty (Pfizer/BioNTech) vaccine
  * First dose or complete cycle of Spikevax (Moderna) vaccine
  * First dose or complete cycle of AstraZeneca/Vaxzevria vaccine
  * Complete cycle of vaccination using one type of vaccine for the first dose and a different type for the second dose
  * Janssen (Johnson & Johnson) vaccine (single dose)

SUMMARY:
Covid-19 vaccines offered a good opportunity to counteract the spread of Sars-Cov-2 infection among the general population, reducing significantly both morbidity and mortality.

Nevertheless, after the first and second doses of vaccination (regardless of the type of vaccine used) several women required gynaecological visits claiming menstrual Irregularities or abnormal uterine bleeding. Considering this anecdotal evidence, a questionnaire was designed to investigate systematically whether menstrual Irregularities or abnormal uterine bleeding occurred in a significant percentage of women undergoing first and second doses of covid-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent first dose or complete cycle of covid-19 vaccine, regardless of the type of vaccine used.

Exclusion Criteria:

* Women undergoing any kind of hormonal therapy, including combined oral contraceptives, oral/vaginal progestins, intrauterine devices, GnRH-analogues, aromatase inhibitors, hormonal replacement therapy in menopause;
* Surgical menopause (hysterectomy and/or bilateral oophorectomy);
* Breastfeeding.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who underwent first dose or complete cycle of covid-19 vaccine, regardless of the type of vaccine used.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Frequency of the menstrual cycle | 30 days after the administration of the first and second doses of vaccine
  In women of reproductive age, any frequency shorter than 25 days or longer than 36 days will be defined as abnormal
Quantity of the menstrual cycle | 30 days after the administration of the first and second doses of vaccine
  In women of reproductive age, any quantity less than 30 ml or more than 80 ml will be defined as abnormal
Duration of the menstrual cycle | 30 days after the administration of the first and second doses of vaccine
  In women of reproductive age, any duration shorter than 3 days or longer than 7 days will be defined as abnormal

SECONDARY OUTCOMES:
Post-menopausal bleeding | 30 days after the administration of the first and second doses of vaccine
  Any bleeding occurred in post-menopausal women

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Ph.D., Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- University of Insubria, Varese, Italy